CLINICAL TRIAL: NCT02703285
Title: Are Medical Personnel Can Correctly Recognize the Chest Sounds?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Lukasz Szarpak, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02.013.1MR
Record Dates: First submitted 2016-02-22; First posted 2016-03-09 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Respiration, Artificial
MeSH Terms: conditions — Respiratory Aspiration | interventions — Sound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- questionnaire (Experimental): task of the participants in the study to determine the chest sound based on specific sounds
  Interventions: Other: Sound

INTERVENTIONS:
Other: Sound — task of the participants in the study to determine the chest sound based on specific sounds: Vesicular - Diminished; Expiratory Wheeze; Bronchovesicular; pneumonia; pulmonary Oedema; Stridor; Agonal respiration

SUMMARY:
The study aims to validate the interpretation of breath sounds by medical personnel

DETAILED DESCRIPTION:
task of the participants in the study to determine the chest sound based on specific sounds

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* paramedics, nurses, physicians

Exclusion Criteria:

* not meet the above criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
breathing sounds measured by questionnaire | 1 day
  study participants selective listening to breath sounds, must mark in questionnaire what is the type of sound. 8 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided